CLINICAL TRIAL: NCT03304093
Title: Immunotherapy by Nivolumab After Prior Chemotherapy for HIV+ Patients With Advanced Non-small Cell Lung Cancer (NSCLC): IFCT-CHIVA2 Phase IIa Trial
Brief Title: Immunotherapy by Nivolumab for HIV+ Patients
Acronym: CHIVA2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1602
Record Dates: First submitted 2017-09-19; First posted 2017-10-06 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-03

CONDITIONS: Non Small Cell Lung Cancer Metastatic; Non Small Cell Lung Cancer Stage IIIB; HIV/AIDS
Keywords: IFCT; VIH; Nivolumab; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Acquired Immunodeficiency Syndrome | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab 3mg/kg every 2 weeks
  Interventions: Drug: Nivolumab Injection

INTERVENTIONS:
Drug: Nivolumab Injection — Nivolumab 3mg/kg every 2 weeks

SUMMARY:
Two Phase III trials showed superiority in terms of efficacy and tolerance of nivolumab in second-line treatment compared to docetaxel in metastatic NSCLC in the general population, so it is important to evaluate this treatment in PLWHIV (Patient Living With HIV) in maximum security conditions, taking into account their specificities and complex underlying immunological status. As NSCLC in PLWHIV is a rare tumour, a phase 2 trial, using DCR (Disease Control Rate) data, would be able to recruit a sufficient number of patients, in a reasonable period of time, to provide a proof of concept of the safety and efficacy of nivolumab in this population. Therefore, we think that an open-label, one arm phase 2 trial, with a rapid accrual, would be currently a crucial approach and a window of opportunity to explore whether nivolumab could find its place in PLWHIV with NSCLC. Such a trial is typically a trial for an academic sponsor, experienced in PLWHIV with NSCLC, which previously showed its ability to recruit patients with such a rare disease as the IFCT did with the IFCT-1001 CHIVA trial, testing carboplatin plus pemetrexed followed by pemetrexed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. HIV1 or HIV2, regardless of CD4 cell count
3. HIV Viral load <200 copies/mL
4. Proven histologically and/or cytologically, stage IIIB-IV or metastatic relapse post-surgery non-small cell lung cancer (NSCLC)
5. Disease recurrence or progression during/after at least one prior platinum doublet-based chemotherapy regimen for advanced or metastatic disease
6. Measurable disease by Computed tomography (CT)/Magnetic resonance imaging (MRI) per RECIST 1.1 criteria
7. Performance status (PS) 0, 1 or 2
8. Written informed consent
9. Patients must have adequate organ function: creatinine clearance > 40 mL/min (Cockcroft, MDRD or CKD-Epi formula or 24h Urine Calculate creatinine clearance from a 24h urine collection ), neutrophiles count > 1500/mm3; platelets > 100 000/mm3 ; hemoglobin > 9 g/dL; hepatic enzymes < 3N with total bilirubin ≤ 1.5 × ULN (upper limit of normal) except subjects with documented Gilbert's syndrome (≤ 5 × ULN) or liver metastasis, who must have a baseline total bilirubin ≤ 3.0 mg/dL
10. Patients must receive appropriate care and treatment for HIV infection including ART when clinically indicated and subjects should be under the care of a physician experienced in HIV management. In case of recent introduction of cART and CD4 levels <50 cells/ml, inclusion will be possible provided subjects had at least 4 weeks of treatment prior to inclusion, to avoid clinical type IRIS (immune inflammatory syndrome reconstitution). All antiretroviral treatments are allowed.
11. Females of childbearing potential who are sexually active with a nonsterilized male partner must use a highly effective method of contraception for 28 days prior to the first dose of investigational product, and must agree to continue using such precautions for 6 months after the final dose of investigational product; cessation of contraception after this point should be discussed with the referent physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. They must also refrain from egg cell donation for 6 months after the final dose of investigational product. Men receiving nivolumab and who are sexually active with women of childbearing potential will be instructed to adhere to contraception (appendix I) for a period of 31 weeks after the last dose of nivolumab.
12. Persons deprived of liberty could be eligible because the expected benefice (improvement of disease control rate) justifies the foreseeable risk (adverse reaction of nivolumab).

Exclusion Criteria:

1. Concurrent malignancies requiring active intervention
2. Active Infection
3. Patient with known EGFR activating tumor mutation or known ALK or ROS1 gene rearrangement not treated with the appropriate targeted therapy.
4. History of immunological events related to HIV: lymphoid interstitial pneumonitis (LIP), non-infectious uveitis, encephalitis and other manifestations of CD8 lymphocyte infiltration syndrome, HIV-associated nephropathy (HIVAN).
5. Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
6. Active or history of inflammatory bowel disease (eg, diverticulitis, colitis, Crohn's, coeliac disease or other serious gastrointestinal chronic conditions associated with diarrhea). Note that diverticulosis is permitted.
7. Symptomatic cerebral metastasis unless treated by brain radiotherapy which will be completed for at least 15 days before the beginning of the treatment; subjects with carcinomatous meningitis.
8. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
9. The last dose of prior chemotherapy or radiation therapy (with the exception of palliative radiotherapy) was received less than 3 weeks prior to inclusion;
10. History of primary immunodeficiency, history of organ transplant that requires therapeutic immunosuppression and the use of immunosuppressive agents within 28 days of inclusion or a prior history of severe (grade 3 or 4) immune mediated toxicity from other immune therapy.
11. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of inclusion. Intranasal/inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
12. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control.
13. Legally protected adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate | 8 weeks

SECONDARY OUTCOMES:
Progression Free Survival | 6 months and one year
  Time between the date of inclusion and the first date of documented progression or death due to any cause, whichever occurs first. Subjects who die without a reported progression will be considered to have progressed on the date of their death. Subjects who did not progress or die will be censored on the date of their last evaluable tumor assessment.
Overall Survival | 6 months and one year
  Time elapsed between the date of inclusion and death. Subjects who did not die will be censored on the last date a subject was known to be alive.
Tolerance | 8 weeks, 6 months and one year
  Adverse Events (AEs) grade (NCI-CTC 4.0)
Responses rate according to tissue PD-L1 expression | 8 weeks
Quality of life measured by LCSS questionnaire | After 2, 3, 5, 7 and 9 cycles (each cycle is 14 days)
Duration of response | 8 weeks, 6 months and one year
impact on HIV control and immunological, other associated chronic infection susceptible of reactivation and potential occurrence of autoimmunity | 8 weeks, 6 months and one year

OTHER OUTCOMES:
Monitor HIV, CMV, EBV, HBV, HCV, HHV-8-specific T cell responses in PBMC | Cycle 1, 2, 3, 9, 15, 27, 51 and end of treatment (each cycle is 14 days)
Monitor the HIV reservoirs (HIV-DNA) and the residual HIV replication as well as EBV CMV, HBV, HCV, HHV-8 viral load | Cycle 1, 2, 3, 9, 15, 27, 51 and end of treatment (each cycle is 14 days)
Monitor T cell activation/ exhaustion/differentiation and immune check point expression | Cycle 1, 2, 3, 9, 15, 27, 51 and end of treatment (each cycle is 14 days)
Description of gene mutation that appear to be crucial for the response to immunotherapy or for adverse effects of immunotherapy | Cycle 1, 2, 3, 9, 15, 27, 51 and end of treatment (each cycle is 14 days)
Immune monitoring of adverse effects | Cycle 1, 2, 3, 9, 15, 27, 51 and end of treatment (each cycle is 14 days)
Describe the tumoral microenvironment of NSCLC before nivolumab exposure (CD4, CD8, CD3 infiltrate, PD-1, PD-L1 expression) | At enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Armelle LAVOLE, MD, Principal Investigator — APHP Hôpital Tenon; Jacques CADRANEL, MD, PhD, Principal Investigator — APHP Hôpital Tenon
Locations (18):
- France (18):
  - CH d'Avignon, Avignon
  - CH de la Côte Basque, Bayonne
  - CH Cahors, Cahors
  - CH, Colmar
  - CHI Créteil, Créteil
  - Centre Hospitalier - Pneumologie, Le Mans
  - Hôpital de la Croix Rousse, Lyon
  - AP-HM Hôpital Nord, Marseille
  - Montpellier - CHRU, Montpellier
  - Montpellier - ICM, Montpellier
  - APHP - Hopital Tenon - Pneumologie, Paris
  - Paris - APHP Bichat, Paris
  - Paris - Pitié-salpêtrière, Paris
  - CH de Pau, Pau
  - Saint Brieuc - CHG, Saint-Brieuc
  - NHC - Pneumologie, Strasbourg
  - Suresnes - Hopital Foch, Suresnes
  - CHU Toulouse - Pneumologie, Toulouse

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT03304093/Prot_000.pdf